CLINICAL TRIAL: NCT01405235
Title: A Prospective, Randomized Phase III Study to Compare the Effects of Paclitaxel and Topotecan to Those of Cisplatin and Topotecan for Treatment of Patients With Recurrent and Persistent Cervical Cancer
Brief Title: Study on Paclitaxel Plus Topotecan in Comparison With Topotecan Plus Cisplatin in Recurrent or Persistent Cervical Carcinoma
Acronym: AGO-Zervix-1
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut fuer Frauengesundheit (Other)
Collaborators: GlaxoSmithKline (Industry); Schantl Pharma Service, Germany (Unknown)
Responsible Party: Frau Dr. med. Patricia Oppelt, Institut fuer Frauengesundheit GmbH
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IFG-01-0106
Record Dates: First submitted 2011-07-27; First posted 2011-07-29 (Estimated); Last update posted 2012-04-12 (Estimated); Status verified 2006-09

CONDITIONS: Recurrent, Persistent or Metastasized Cervical Cancer
Keywords: Paclitaxel/Topotecan; Cisplatin/Topotecan
MeSH Terms: conditions — Recurrence | interventions — Paclitaxel; TP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm B: Cisplatin/Topotecane (Active Comparator): Topotecan 0.75 mg/m2/d i.v. on Days 1- 3 in combination with Cisplatin 50 mg/m2 i.v. on Day 1, q 21 d
  Interventions: Drug: Cisplatin/Paclitaxel
- Arm A: Paclitaxel/Topotecan (Experimental): Paclitaxel 70 mg/m2/d i.v. on Days 1, 8, and 15 in combination with Topotecan 1.75 mg/m2/d i.v. on Days 1, 8, and 15, q 28 d
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel 70 mg/m2/d i.v. on Days 1, 8, and 15 in combination with Topotecan 1.75 mg/m2/d i.v. on Days 1, 8, and 15, q 28 d
  Arms: Arm A: Paclitaxel/Topotecan
Drug: Cisplatin/Paclitaxel — Topotecan 0.75 mg/m2/d i.v. on Days 1- 3 in combination with Cisplatin 50 mg/m2 i.v. on Day 1, q 21 d
  Arms: Arm B: Cisplatin/Topotecane

SUMMARY:
Current planning for studies involving patients with recurrent, persistent, or metastasized cervical cancer must take into consideration that up to 75% of all patients are assumed to have already been treated with cisplatin in conjunction with radiation therapy. It seems questionable to continue to treat patients with cisplatin when cancer has recurred. Thus, it is important to seek alternative active combinations. The studies GOG 169 and 179 demonstrated that a combination of paclitaxel and cisplatin was superior to a cisplatin monotherapy with respect to therapeutic response and progression-free survival, as was a combination of topotecan and cisplatin with respect to therapeutic response, progression-free survival, and total survival. To achieve further improvement in total survival and to answer questions regarding the value of using a platinum-free combination, we propose that a study should be conducted to compare the efficacy of a platinum-free combination of paclitaxel and topotecan to a combination of cisplatin and topotecan.

DETAILED DESCRIPTION:
Design: This will be a prospective, randomized, multicenter, non-blinded phase III A study.

Dosages: Arm A Paclitaxel 70 mg/m2/d i.v. on Days 1, 8, and 15 in combination with Topotecan 1.75 mg/m2/d i.v. on Days 1, 8, and 15, q 28 d Arm B Topotecan 0.75 mg/m2/d i.v. on Days 1- 3 in combination with Cisplatin 50 mg/m2 i.v. on Day 1, q 21 d Duration of Therapy: Each patient will participate in the study until a maximum of six cycles have been completed, or until there is evidence of disease progression, or until toxicity prevents further therapy. Patients with continued response or stable disease may continue to participate in the study for an additional 3 cycles beyond the original 6 cycles with consent of the Study Director, but this must be documented in the CRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed recurrent, persistent, or metastasized squamous cell carcinoma, adenosquamous carcinoma, or adenocarcinoma of the cervix, for which a curative treatment by operation and/or radiation therapy is not possible.
* Patients must have been previously treated with cisplatin in the context of radiochemotherapy.
* All patients must present with measurable disease. Measurable disease is defined as a minimum of one lesion that can be accurately measured in at least one dimension (longest dimension to be recorded). Each lesion must measure ≥ 20 mm when measured by conventional techniques, including palpation, x-ray, CT, and MRI, or ≥ 10 mm when measured by spiral CT. Patients must have at least one "target lesion" that can be used to evaluate response according to RECIST criteria during this study.
* When a biopsy is performed, it should be performed on this lesion. A lesion outside of the irradiated area should ideally be selected as the "target lesion" on patients who have tumors both inside and outside a previously irradiated area. A previously irradiated lesion may only be considered as a "target lesion" if, after the radiation therapy had been completed, this lesion objectively led to a diagnosis of recurrence, or progress specific to this lesion was observed.
* Patients must display the following:

  * Sufficient hematologic function: absolute neutrophil count ≥ 1.
  * 500/μl; granulocytes > 3,000/μl; thrombocytes ≥ 100,000/μl.
  * Sufficient renal function: serum creatinine ≤ 1.2 mg/dl. In patients with a serum A prospective, randomized phase III study to compare the effects of Paclitaxel and Topotecan to those of Cisplatin and Topotecan for treatment of patients with recurrent or persistent cervical cancer Page 24 Study Protocol Version 1.1 dated 09/25/2006 creatinine of > 1.2 mg/dl, the results of a 24-hour creatinine clearance must yield a level > 50 cm3/min for eligibility.
  * Sufficient liver function: bilirubin ≤ 1.5 times the institutional upper limit of normal, GOT, alkaline phosphatase ≤ 3 times the institutional upper limit of normal.
  * Patients must display an ECOG performance status of 0-2 (Karnofsky > 60%).
  * Patients must have recovered from the aftereffects of any surgery, radiation therapy, or chemotherapy. A minimum of six weeks must have passed since the last administration of chemotherapy, and at least three weeks must have passed since the last treatment with radiation alone.
  * Patients must have signed an official consent document which also authorizes the release of personal health information. Patients unable to give their consent independently may not participate in the study.
  * Patients must fulfill all the requirements defined in Section 8.1, including completion of a baseline quality of life questionnaire, prior to their inclusion in the study.
  * Patients must be free of clinically significant infection.
  * Patients must be 18 years of age or older.

Exclusion Criteria:

* Patients with bilateral hydronephrosis which cannot be alleviated by ureteral stents or percutaneous drainage. Patients with a serum creatinine > 1.2 mg/dl but < 1.5 mg/dl and a 24-hour creatinine clearance result of < 50 cm3/min. Patients with a serum creatinine ≥ 1.5 mg/dl. A prospective, randomized phase III study to compare the effects of Paclitaxel and Topotecan to those of Cisplatin and Topotecan for treatment of patients with recurrent or persistent cervical cancer Study Protocol Version 1.1 dated 09/25/2006 Page 25

  * Patients who have received prior chemotherapy, unless the chemotherapy was administered with concomitant radiation therapy.
  * Patients who are pregnant or lactating.
  * Patients with craniospinal metastases.
  * Patients with a concomitant malignant disease, with the exception of nonmelanoma skin cancer.
  * Patients with a previous invasive malignant disease (other than nonmelanoma skin cancer) showing evidence of this disease within the last 5 years, or for whom the therapy to be administered during this study is contraindicated due to previous treatment received for this malignant disease.
  * Patients who are participating in another clinical study at the same time or who will have done so up to 30 days before the planned end of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2006-09; Primary Completion 2012-06 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Changes in target lesion according to RECIST 1.0 | week 12

CONTACTS AND LOCATIONS:
Overall Officials: Falk Thiel, Dr. med., Study Chair — Frauenklinik Universitätsklinikum Erlangen
Locations (1):
- Universitätsfrauenklinik, Erlangen, Bavaria, Germany

REFERENCES:
- [Derived] Gass P, Thiel FC, Haberle L, Ackermann S, Theuser AK, Hummel N, Boehm S, Kimmig R, Reinthaller A, Becker S, Hilpert F, Janni W, Vergote I, Harter P, Emons J, Hein A, Beckmann MW, Fasching PA, Poschke P; AGO Uterus Commission. Primary results of the AGO-Zervix-1 Study: A prospective, randomized phase III study to compare the effects of paclitaxel and topotecan with those of cisplatin and topotecan in the treatment of patients with recurrent and persistent cervical cancer. Gynecol Oncol. 2024 Apr;183:25-32. doi: 10.1016/j.ygyno.2024.03.002. Epub 2024 Mar 14. PMID 38490057